CLINICAL TRIAL: NCT02721771
Title: Acid-base Disturbances and Ultrasound Markers as Biological Predictors of Maternal and Fetal Outcomes in Severe Late Onset Preeclampsia
Brief Title: Acid-Base and Point of Care Ultrasound in Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Medical University of Vienna (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Robert Dyer, Professor Robert Anthony Dyer, University of Cape Town
Other Study IDs: UCapeTown
Record Dates: First submitted 2016-03-10; First posted 2016-03-29 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasound examination — echocardiographic diastology and bilateral B-line pattern will be assessed. Optic nerve sheath diameter will be assessed.
  Other Names: ONSD, B-pattern, diastology

SUMMARY:
Preeclampsia remains a leading cause of maternal morbidity and mortality, in both the developed and developing world. It is a complex, multisystem disease which, in its severe form, affects the cardiovascular, renal, hepatic, neurological and haematological systems. The University of Cape Town-associated medical institutions alone were responsible for the treatment of 800 women in 2014, who were classified as having preeclampsia with severe features. Given the complexity of the disease, anesthetic management for Caesarean section in these patients remains very challenging.

Recent studies have begun to demonstrate novel markers of preeclampsia severity, including point-of-care ultrasound (POC-US) and acid-base (AB) abnormalities. For example, pilot studies have demonstrated that approximately 25% of women diagnosed with severe preeclampsia show signs of increased intracranial pressure and elevated lung water as evaluated by point of care ultrasound. These findings could serve as noninvasive markers of disease severity, and thus may be used to predict maternal and fetal outcome in preeclamptic women. Point of care ultrasound is playing an increasing role in perioperative diagnosis, and newer, less expensive devices are continuously being developed, and will in all likelihood play an important role in South Africa in the near future.

In a recent trial performed at the University of Cape Town, a comprehensive acid-base analysis in severe preeclamptic women demonstrated significant abnormalities in independent acid-base determinants. In addition, strong indications were found that changes in acid-base status in preeclampsia are more pronounced earlier in pregnancy and are associated with urgent deliveries. As in other clinical arenas in critically ill patients, acid-base abnormalities are associated with increased lung water, increased intracranial pressure, and outcome, and we hypothesize that similar associations might be found in severe preeclamptic women. Therefore, one aim of this study is to evaluate the association of venous acid base abnormalities (an inexpensive and readily available test) observed in late onset severe preeclampsia and organ manifestations identified with ultrasound, a well-validated and robust tool for identifying these manifestations. Investigators will further examine the association between ultrasound findings and/or venous acid-base abnormalities with urgent delivery. It is intended to do a subsequent comparison between early- and late onset preeclampsia, when a suitable tertiary site has been identified.

DETAILED DESCRIPTION:
I. Introduction / Specific Aims Preeclampsia is a major cause of maternal mortality (15-20 % in developed countries) and acute and long-term morbidity for the mother and newborn. It is a multi-system disorder characterised by abnormal vascular response to placentation, associated with increased systemic vascular resistance, enhanced platelet aggregation, activation of the coagulation system, and endothelial dysfunction. Preeclampsia is defined by a number of signs and symptoms, but is characterized by multi-organ changes that encompass the central nervous system (CNS), lungs, liver, kidneys, systemic vasculature, coagulation, and the heart .

Derived from other clinical arenas of intensive care medicine, new potential markers of disease severity in women diagnosed with preeclampsia have recently been identified. Using noninvasive point-of-care (POC) ultrasound, pulmonary interstitial edema and raised intracranial pressure were identified in 25% and 20% respectively of women showing features of severe preeclampsia. In addition, echocardiographic and laboratory studies in women diagnosed with preeclampsia indicate an incidence of diastolic dysfunction and increased left ventricular end-diastolic pressure (LVEDP) in up to 30%. These findings could have a significant impact on maternal outcome and the detailed methodology of anesthesia care for the parturient with severe preeclampsia (PreE), including the mode of anesthesia, positioning of the patient, fluid management, and hemodynamic goals.

In a recent investigation performing a comprehensive physicochemical acid/base analysis in pre-eclamptic women (AB-PreE-Trial), the presence of simultaneous hypoalbuminaemic alkalosis and hyperchloraemic acidosis was identified. In addition, investigators found indications that hypoalbuminaemic alkalosis is more marked in early versus late onset disease and is associated with mode of delivery. In other critical care arenas it has been shown that reduced albumin and acid-base abnormalities are associated with pulmonary interstitial edema, elevated intracranial pressure (ICP), and poor clinical outcomes. Venous acid-base analysis may therefore be a widely available and inexpensive marker of pulmonary interstitial edema and elevated ICP in preeclampsia, with potentially important impact on anesthesia care. Therefore, one aim is to evaluate the association between elevated base excess to changes in albumin concentration (BE(Alb)) with pulmonary interstitial edema and increased ICP (both evaluated with non-invasive ultrasound) in patients with late onset severe preeclampsia. Investigators will further evaluate for an association with urgent delivery (fetal or maternal indication).

Long-term goal will be to use findings to guide clinical decision-making by anaesthetists to identify individual patients with acute organ system failures, helping better plan anaesthetic management during Cesarean delivery. Also, the findings from a larger future study could predict maternal and fetal complications, and show differences between early- and late onset disease. This should be of significant future benefit in the South African context, where preeclampsia is a leading cause of maternal morbidity and mortality.

II. Aims

Aim 1: To explore the association between ultrasound findings and/or venous acid-base abnormalities, with urgent delivery.

It is hypothesised that patients with acid-base changes secondary to albumin, interstitial edema and/or elevated ICP will experience a greater proportion of urgent deliveries, compared to patients without these abnormalities.

Aim 2: To determine the association between pulmonary interstitial edema and increased ICP with changes in BE(Alb).

Primary Hypothesis: Based on prior studies showing the association of low albumin with increased extravascular lung water and worse cerebral edema it is hypothesised that the mean BE(Alb) will be higher in patients with pulmonary interstitial edema and increased ICP (assessed with POC ultrasound), compared to patients without interstitial edema and normal ICP. Point-of-care ultrasound is a validated method of identifying both pulmonary interstitial edema and elevated ICP.

Sample size calculations:

Aim 1: Among patients with late onset disease, prior data suggests that 30% of patients will have a BE(Alb) > 4 meq/L, with a rate of fetal distress >70% in this population, as compared to a fetal distress rate of 25% in women with a BE(Alb) < 4 meq/L. Based on the observation that 70% of women in late onset disease will have a BE(Alb) < 4 meq/L at diagnosis, and considering an alpha level of 0.05 and power of 0.8, 70 patients will be needed to reject null hypothesis of predicting delivery status with BE(alb) > 4mEq/L.

Aim 2: In addition, available data suggests that the incidence of elevated intracranial pressure and interstitial pulmonary edema diagnosed by ultrasound in severe preeclampsia is approximately 25%, and an elevated BE (Alb) is found in approximately 30% of patients with severe preeclampsia. Prior data in critically ill patients indicates a mean albumin of 2.8 g/dL (SD 0.7) in patients with normal lung water, compared a mean albumin of 2.2 g/dL (SD 0.7) in patients with increased lung water. When converted to the BE (Alb) scale (assuming a mean pH of 7.4) and with the biologically plausible assumption of a similar relationship with ICP, in order to show a statistically meaningful difference in the mean BE (Alb) level among patients with severe preeclampsia with and without interstitial edema and with and without elevated ICP, we will need to recruit a total of 80 patients, with an alpha level of 0.05 and a power of 0.9. Furthermore, on the BE (Alb) scale, the mean BE (Alb) of the low albumin group (mean albumin of 2.2 g/dL) is approximately equal to a BE (Alb) of 4 meq/L and may represent an important clinical endpoint. Thus, assuming a normal distribution, 50% of this group is expected to have a BE (Alb) > 4 meq/L. The increased albumin group (mean albumin of 2.8 g/dL) lies approximately 1 standard deviation from the decreased albumin group, and assuming a normal distribution, we would expect 18% of this group to exceed the BE (Alb) > 4 meq/L cut point. Using these two proportions, a chi-squared test with a sample ratio of 3:1, power of 0.8, and alpha level of 0.05 will require a total sample size of 84 patients (21 with the ultrasound findings and 63 without findings).

ELIGIBILITY:
Inclusion Criteria:

* age > 18years
* previously healthy
* new late onset severe preeclampsia

Exclusion Criteria:

* labour
* chronic obstructive pulmonary disease (COPD)
* collagen disorder
* ho lithium intoxication
* ho of methanol, ethanol, salicylates ingestion
* HIV
* regular ingestion of antacids
* chronic renal disease
* chronic hepatic disease
* urinary tract infection (UTI),
* infection, sepsis
* BMI>50
* acute asthma
* unable to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with late onset severe preeclampsia according to the definition of the Royal college of obstetricians and gynaecologists.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Association BE(alb) and with delivery outcome | 24hours
  Comparison number of patients with abnormal BE(alb) with number of patients undergoing emergency cesarean section (indicated through abnormal CTG).
Correlation BE(alb) with comet score and optic nerve sheath diameter (ONSD) | 24hrs
  correlation BE(alb) with comet score and optic nerve sheath diameter (ONSD)

SECONDARY OUTCOMES:
Association B-pattern on lung ultrasound and delivery outcome | 24hrs
  Comparison number of patients with B-pattern on lung ultrasound with number of patients undergoing emergency cesarean section (indicated through abnormal CTG).
Association increased intracranial pressure (ICP) based on ONSD and delivery outcome | 24hrs
  Comparison number of patients with increased ICP (=ONSD>5.8mm) with number of patients undergoing emergency cesarean section (indicated through abnormal CTG).

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Dyer, MD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape/Observatory, South Africa

REFERENCES:
- [Derived] Ortner CM, Krishnamoorthy V, Neethling E, Flint M, Swanevelder JL, Lombard C, Fawcus S, Dyer RA. Point-of-Care Ultrasound Abnormalities in Late-Onset Severe Preeclampsia: Prevalence and Association With Serum Albumin and Brain Natriuretic Peptide. Anesth Analg. 2019 Jun;128(6):1208-1216. doi: 10.1213/ANE.0000000000003759. PMID 31094790